CLINICAL TRIAL: NCT07103993
Title: Food Intake and Thermogenesis in High Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Gary Farkas, Assistant Professor, University of Miami
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: 20250335
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: SCI - Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low meal condition group (Experimental): Subjects will be in this group for up to 3 weeks.
  Interventions: Other: Low meal condition; Other: Ad-libitum control condition
- Moderate meal condition group (Experimental): Subjects will be in this group for up to 3 weeks.
  Interventions: Other: Moderate meal condition; Other: Ad-libitum control condition
- High meal condition group (Experimental): Subjects will be in this group for up to 3 weeks.
  Interventions: Other: High meal condition; Other: Ad-libitum control condition

INTERVENTIONS:
Other: Low meal condition — Participants will consume a standardized meal (500 grams) with a low nutrient modification one time at one visit. Participants will attend one visit per week for 3 weeks. Each is visit separated by one week and each visit will take approximately 6 hours
  Arms: Low meal condition group
Other: Moderate meal condition — Participants will consume a standardized meal (500 grams) with a moderate nutrient modification one time at one visit. Participants will attend one visit per week for 3 weeks. Each is visit separated by one week and each visit will take approximately 6 hours.
  Arms: Moderate meal condition group
Other: High meal condition — Participants will consume a standardized meal (500 grams) with a high nutrient modification one time at one visit. Participants will attend one visit per week for 3 weeks. Each is visit separated by one week and each visit will take approximately 6 hours.
  Arms: High meal condition group
Other: Ad-libitum control condition — The ad-libitum meal consists of 600-700 g of a standardized control meal one time at all visits. Participants will attend one visit per week for 3 weeks. Each visit is separated by one week and each visit will take approximately 6 hours.

SUMMARY:
The purpose of this research is to determine the effects of food on cardiovascular and metabolic health in men with and without spinal cord injury (SCI).

ELIGIBILITY:
Inclusion Criteria:

SCI and Controls

* Men
* Physically inactive (<150 minutes per week of moderate-vigorous activity intensity for the preceding 3 months)
* Weight stable: body mass ±3 kilograms (kg) for past 3 months

SCI Only

* Chronic SCI (≥ 1-year post-injury)
* Motor-complete SCI American Spinal Injury Association Impairment Scale (AIS) A and B
* T6 injuries and above that can independently feed themselves

Exclusion Criteria:

SCI and Controls

* Uncompensated thyroid disease
* Diabetes
* Swallowing or gastrointestinal pathologies
* Allergies or aversions to foods/ingredients
* Prescribed prokinetic, antipsychotic, or anti-obesity agents

SCI Only

* Incomplete SCI AIS C or D
* Ventilator-dependent

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male subjects
Enrollment: 56 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Diet induced thermogenesis (DIT) | up to 3 weeks (collected during each of the intervention visits)
  Diet-induced thermogenesis (DIT) will be measured using indirect calorimetry. A portable mask-based metabolic system, which will measure expired air to calculate dietary-induced thermogenesis defined as the energy expended above resting and the proportion of meal energy expended postprandially (postprandial kilocalorie (kcal) expended/total meal kcal) where a higher value means more energy is expended.
Hunger Series Visual Analog Scale | up to 3 weeks (collected during each of the intervention visits)
  Satiety will be measured using the Hunger Series Visual Analog Scale (HSVAS), which assesses subjective appetite. Each scale is defined at 0 as "not at all hungry" and 100 as "totally/a lot/very hungry". A sum score will be calculated.
Post ad-libitum energy intake measured in grams | up to 3 weeks (collected during each of the intervention visits)
  This value will be expressed as a ratio of energy consumed to energy requirements (energy intake/energy requirements x 100) and will be recorded in grams.

CONTACTS AND LOCATIONS:
Overall Officials: Gary J Farkas, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami - Miami Project to Cure Paralysis, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No